CLINICAL TRIAL: NCT04772313
Title: A Phase 4, Multicenter, Open-label, Efficacy and Safety Trial of Pegloticase and Methotrexate Co-administered in Patients With Uncontrolled Gout Who Have Previously Received Pegloticase Monotherapy But Did Not Maintain a Serum Uric Acid Response
Brief Title: Pegloticase and Methotrexate Co-administered in Participants With Uncontrolled Gout Who Previously Failed Pegloticase Monotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZNP-KRY-407
Record Dates: First submitted 2021-02-24; First posted 2021-02-26 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Uncontrolled Gout
Keywords: Gout
MeSH Terms: conditions — Gout | interventions — Pegloticase; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pegloticase plus Methotrexate (MTX) (Experimental): Pegloticase (8 mg) intravenous (IV) every two weeks. Methotrexate (15 or 25 mg weekly) SC.
  Interventions: Biological: Pegloticase; Drug: Methotrexate (MTX)

INTERVENTIONS:
Biological: Pegloticase — Participants will receive pegloticase with MTX for up to 24 weeks during the treatment period. Participants may opt to receive pegloticase with MTX for an additional 24 weeks.
Drug: Methotrexate (MTX) — Participants will receive MTX during the run-in period then pegloticase with MTX for up to 24 weeks during the treatment period. Participants may opt to receive pegloticase with MTX for an additional 24 weeks.

SUMMARY:
This is a Phase 4, multicenter, open-label trial of pegloticase with methotrexate (MTX) in adult participants with uncontrolled gout who were previously treated with pegloticase without a concomitant immunomodulator and stopped pegloticase due to failure to maintain serum uric acid (sUA) response and/or a clinically mild infusion reaction (IR). Approximately 30 participants will be enrolled. Pegloticase + MTX will be administered for approximately 24 weeks, with an optional extension up to 48 weeks.

The trial design will include 5 distinct components:

1. Screening Period, lasting up to 42 days;
2. 6-week MTX Tolerability Assessment Period (hereafter referred to as the MTX Run-in Period);
3. 24-week Pegloticase + MTX Treatment Period, which will include a Week 24/End of Trial/Early Termination Visit (subjects that end MTX and pegloticase treatment prior to the Week 24 will remain on trial for follow up until the Week 24 visit)
4. Optional Pegloticase + MTX Extension Period up to 24 weeks
5. 30-Day Post Treatment Follow -up

DETAILED DESCRIPTION:
All participants who meet eligibility criteria at Screening will begin once-weekly subcutaneous (SC) MTX Run-in period. Participants must be able to tolerate MTX at a minimum dose of 15 mg during the 6-week MTX Run-in Period to be eligible to participate in the Pegloticase + MTX Treatment Period.

All participants who meet the inclusion/exclusion criteria and complete the MTX Run-in Period will be considered enrolled participants. During the Pegloticase + MTX Treatment Period, pegloticase 8 mg will be administered IV every 2 weeks and MTX SC weekly.

Two sequential cohorts of participants will be enrolled in this trial. Cohort 1 is targeted to enroll 10 participants who previously failed to maintain sUA response with pegloticase monotherapy and stopped pegloticase treatment without a history of pegloticase-related infusion reaction.

If the safety assessment during Cohort 1 indicates that the pegloticase infusions are well tolerated, then the trial can begin enrolling Cohort 2 for 20 participants who failed to maintain sUA response with pegloticase monotherapy with or without a history of pegloticase-related clinically mild IRs.

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give informed consent.
2. Willing and able to comply with the prescribed treatment protocol and evaluations for the duration of the trial.
3. Adult men or women ≥18 years of age.
4. Uncontrolled gout, defined by the following criteria:

   * Hyperuricemia during the Screening Period, defined as sUA ≥6 mg/dL, and;
   * Failure to maintain normalization of sUA with xanthine oxidase inhibitors at the maximum medically appropriate dose or with a contraindication to xanthine oxidase inhibitor therapy based on medical record review or subject interview, and;
   * Symptoms of gout, including at least 1 of the following:

     * Presence of at least 1 tophus
     * Recurrent flares, defined as 2 or more flares in the 12 months prior to Screening
     * Presence of chronic gouty arthritis
5. Subject was previously treated with pegloticase without concomitant immunomodulation and stopped pegloticase due to failure to maintain sUA reduction response (had ≥1 sUA >6 mg/dL within 2 weeks post pegloticase infusion) and did not experience an IR (Cohort 1) and/or stopped pegloticase treatment due to pegloticase-related clinically mild IR (Cohort 2).
6. Subject for whom the last pegloticase infusion occurred >6 months prior to Screening.
7. Willing to discontinue any oral urate-lowering therapy for at least 7 days prior to Day 1 and remain off other urate-lowering therapy during the Pegloticase + MTX Treatment Period.
8. Women of childbearing potential (including those with an onset of menopause <2 years prior to Screening, non-therapy-induced amenorrhea for <12 months prior to Screening or not surgically sterile [absence of ovaries and/or uterus]) must have negative serum pregnancy tests during Screening:

   Subjects must agree to use 2 reliable forms of contraception during the trial, 1 of which is recommended to be hormonal, such as an oral contraceptive. Hormonal contraception must be started ≥1 full cycle prior to Week -6 (start of MTX) and continue for 30 days after the last dose of pegloticase, or at least 1 ovulatory cycle after the last dose of MTX (whichever is the longer duration after the last dose of pegloticase). Highly effective contraceptive methods (with a failure rate <1% per year), when used consistently and correctly, include implants, injectables, combined oral contraceptives, some intrauterine devices, sexual abstinence or vasectomized partner.
9. Men who are not vasectomized must agree to use appropriate contraception so as to not impregnate a female partner of reproductive potential during the trial, beginning with the initiation of MTX at Week -6 and continuing for at least 3 months after the last dose of MTX.
10. Able to tolerate MTX at SC doses of at least 15 mg during the MTX Run-in Period, regardless of estimated glomerular filtration rate (eGFR) status.

Exclusion Criteria:

1. Known history of medically confirmed prior anaphylactic reaction.
2. Known history of moderate or severe IR (including but not limited to difficulty in breathing, hypotension, generalized urticaria, generalized erythema, angioedema and/or required treatment with IV steroids or epinephrine; or other serious adverse events (SAEs) related to pegloticase or any other pegylated product treatment.
3. Weight >160 kg (352 pounds) at Screening.
4. Any serious acute bacterial infection, unless treated and completely resolved with antibiotics at least 2 weeks prior to the Week 6 Visit.
5. Severe chronic or recurrent bacterial infections, such as recurrent pneumonia or chronic bronchiectasis.
6. Current or chronic treatment with systemic immunosuppressive agents, such as MTX, azathioprine, cyclosporine, leflunomide, cyclophosphamide or mycophenolate mofetil.
7. Current treatment with prednisone >10 mg/day or equivalent dose of another corticosteroid on a chronic basis (defined as 3 months or longer).
8. Known history of any solid organ transplant surgery requiring maintenance immunosuppressive therapy.
9. Known history of hepatitis B virus surface antigen positivity or hepatitis B DNA positivity, unless treated, viral load is negative and no chronic or active infection confirmed by hepatitis B virus serology.
10. Known history of hepatitis C virus RNA positivity, unless treated and viral load is negative.
11. Known history of human immunodeficiency virus positivity.
12. glucose-6-phosphate dehydrogenase (G6PD) deficiency (tested at the Screening Visit).
13. Severe chronic renal impairment (eGFR <30 mL/min/1.73 m^2) at the Screening Visit based on 4 variable Modification of Diet in Renal Disease [MDRD] formula or currently on dialysis.
14. Non-compensated congestive heart failure, hospitalization for congestive heart failure or treatment for acute coronary syndrome (myocardial infarction or unstable angina) within 3 months of the Screening Visit, current uncontrolled arrhythmia or current uncontrolled blood pressure (>160/100 mm Hg) prior to Week -6.
15. Pregnant, planning to become pregnant, breastfeeding, planning to impregnate female partner, or not on an effective form of birth control, as determined by the Investigator.
16. Prior treatment with another recombinant uricase (rasburicase) or concomitant therapy with a PEG-conjugated drug.
17. Known allergy to pegylated products or history of anaphylactic reaction to a recombinant protein or porcine product.
18. Contraindication to MTX treatment or MTX treatment considered inappropriate.
19. Known intolerance to MTX.
20. Receipt of an investigational drug within 4 weeks or 5 half-lives, whichever is longer, prior to MTX administration at Week -6 or plan to take an investigational drug during the trial.
21. Current liver disease, as determined by alanine transaminase (ALT) or aspartate transaminase (AST) >1.25 × upper limit of normal (ULN) or albumin <lower limit of normal at the Screening Visit.
22. Currently receiving systemic or radiologic treatment for ongoing cancer, excluding nonmelanoma skin cancer.
23. History of malignancy within 5 years other than non-melanoma skin cancer or in situ carcinoma of cervix.
24. White blood cell count <4.0 × 10^9/L, hematocrit <32% or platelet count <75 × 10^9/L.
25. Diagnosis of osteomyelitis.
26. Known history of hypoxanthine-guanine phosphoribosyl-transferase deficiency, such as Lesch-Nyhan and Kelley-Seegmiller syndrome.
27. Unsuitable candidate for the trial (e.g., cognitive impairment), based on the opinion of the Investigator, such that participation might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements or complete the trial.
28. Alcohol use in excess of 3 alcoholic beverages per week.
29. A known intolerance to all protocol standard gout flare prophylaxis regimen (i.e., unable to tolerate any of the following 3 agents: colchicine,nonsteroidal anti-inflammatory drugs (NSAIDs) or low- dose prednisone (≤10 mg/day).
30. Current pulmonary fibrosis, bronchiectasis or interstitial pneumonitis. If deemed necessary by the Investigator, a chest x-ray may be performed during Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2023-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (15):
- United States (15):
  - University of Alabama at Birmingham (UAB) - Center for Education & Research on Therapeutics of Musculoskeletal Disorders, Birmingham, Alabama
  - Arizona Arthritis and Rheumatology Associates, Flagstaff, Arizona
  - Arizona Arthritis and Rheumatology Associates, Glendale, Arizona
  - Arizona Arthritis and Rheumatology Associates, Mesa, Arizona
  - East Bay Rheumatology Medical Group, San Leandro, California
  - Providence St. John's Health Clinic, Santa Monica, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Life Clinical Trials, Margate, Florida
  - IRIS Research and Development, LLC, Plantation, Florida
  - Napa Research, Pompano Beach, Florida
  - GCP Clinical Research, LLC, Tampa, Florida
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Biopharma Informatic, LLC, Houston, Texas
  - Western Washington Arthritis Clinic, Bothell, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants who meet the inclusion/exclusion criteria and completed the MTX Run-in Period were considered enrolled participants and received the first pegloticase infusion on Day 1. Participants who did not complete the MTX Run-in Period were considered screen failures.
Groups:
- Pegloticase Plus Methotrexate: Methotrexate (MTX) 15 or 25 mg subcutaneous (SC) weekly during the 6-week MTX Run-in Period. Pegloticase 8 mg intravenous (IV) every 2 weeks and MTX 15 or 25 mg SC weekly for up to 24 weeks during the treatment period. Participants may opt to receive pegloticase with MTX for an additional 24 weeks.
Period: MTX Run-in Period
Arm/Group | Pegloticase Plus Methotrexate
Started | 13
Completed | 11
Not Completed | 2
Period: Pegloticase + MTX Treatment Period
Arm/Group | Pegloticase Plus Methotrexate
Started | 11
Completed | 5
Not Completed | 6
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 3
Period: Pegloticase + MTX Extension Period
Arm/Group | Pegloticase Plus Methotrexate
Started | 1 (participants continuing in the optional extension period)
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population
Groups:
- Pegloticase Plus Methotrexate: MTX 15 or 25 mg SC weekly during the 6-week MTX Run-in Period. Pegloticase 8 mgIV every 2 weeks and MTX 15 or 25 mg SC weekly for up to 24 weeks during the treatment period. Participants may opt to receive pegloticase with MTX for an additional 24 weeks.
Arm/Group | Pegloticase Plus Methotrexate
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Serum Uric Acid (sUA) Responders (sUA < 6 mg/dL) During Month 6
Description: An sUA responder is defined as a participant achieving and maintaining sUA <6 mg/dL for at least 80% of the time during Month 6 (Weeks 20, 21, 22, 23 and 24).
Time Frame: Month 6
Population: Intent-to-Treat (ITT) Analysis Set: all participants who receive at least 1 dose of pegloticase + methotrexate.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegloticase Plus Methotrexate
Number analyzed (Participants) | 11
percentage of participants | 9.1 [0.2 to 41.3]

2. Secondary Outcome: Percentage of sUA Responders (sUA < 6 mg/dL) During Month 3
Description: An sUA responder is defined as a participant achieving and maintaining sUA <6 mg/dL for at least 80% of the time during Month 3 (Weeks 10 to 14).
Time Frame: Month 3
Population: ITT Analysis Set: all participants who receive at least 1 dose of pegloticase + methotrexate.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegloticase Plus Methotrexate
Number analyzed (Participants) | 11
percentage of participants | 9.1 [0.2 to 41.3]

3. Secondary Outcome: Percentage of Participants Who Experienced Any of the Following Events From Day 1 to Week 24: Infusion Reaction (IR) Leading to Discontinuation of Treatment, Anaphylaxis or Meeting Individual Participant sUA Discontinuation Criteria
Description: Individual participant sUA discontinuation criteria are met when the lowest available interim sUA value after the pegloticase infusion at Week 2, 4, 6, 8, 10 or 12 is less than a 50% reduction from the highest sUA value measured between Screening and pre-infusion on Day 1.
Time Frame: Day1 to Week 24
Population: ITT Analysis Set: all participants who receive at least 1 dose of pegloticase + methotrexate.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegloticase Plus Methotrexate
Number analyzed (Participants) | 11
percentage of participants | 81.8 [48.2 to 97.7]

4. Secondary Outcome: Mean Change From Baseline in Urate Deposition Volume Measured by Dual Energy Computed Tomography (DECT) to Week 24
Description: DECT scans measure urate deposition volume. DECT scans at Week 24 were taken for hands, foot/ankle, and knees.
Time Frame: Baseline to Week 24
Population: ITT Analysis Set: all participants who receive at least 1 dose of pegloticase + methotrexate; participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Pegloticase Plus Methotrexate
Number analyzed (Participants) | 9
cm^3
  Change in Total Urate Volume of Hands: number analyzed (Participants) | 3
  Change in Total Urate Volume of Hands | -0.073 (0.1270)
  Change in Total Urate Volume of Foot/Ankle: number analyzed (Participants) | 3
  Change in Total Urate Volume of Foot/Ankle | -1.540 (1.7545)
  Change in Total Urate Volume of Knees: number analyzed (Participants) | 3
  Change in Total Urate Volume of Knees | -1.207 (0.9073)

5. Secondary Outcome: Mean Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score at Weeks 14 and 24
Description: HAQ-DI is a self-report functional status instrument that is filled out by the participant and measures disability over the past week via 20 questions relating to 8 domains of function: dressing grooming, arising, eating, walking, hygiene, reach, grip, usual activities. For each of the categories, participants reported the amount of difficulty they had in performing 2 or 3 specific subcategory items. The standard disability score is calculated from the 8 categories by dividing the sum of the individual categories by the number of categories answered, yielding a score from 0 (without any difficulty) to 3 (unable to do), with higher values indicating higher disability.
Time Frame: Baseline, Week 14, Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pegloticase Plus Methotrexate
Number analyzed (Participants) | 11
score on a scale
  Change at Week 14: number analyzed (Participants) | 6
  Change at Week 14 | 0.25 (0.617)
  Change at Week 24: number analyzed (Participants) | 5
  Change at Week 24 | 0.10 (0.163)

6. Secondary Outcome: Mean Change From Baseline in Health Assessment Questionnaire (HAQ) Pain Score at Weeks 14 and 24
Description: The HAQ pain scale asks participants to record how much pain they have had in the past week on a scale of 0-100 where zero represents no pain and 100 represents severe pain.
Time Frame: Baseline, Week 14, Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pegloticase Plus Methotrexate
Number analyzed (Participants) | 11
score on a scale
  Change at Week 14: number analyzed (Participants) | 6
  Change at Week 14 | 10.67 (19.664)
  Change at Week 24: number analyzed (Participants) | 5
  Change at Week 24 | -4.00 (15.166)

7. Secondary Outcome: Mean Change From Baseline in HAQ Health Score at Weeks 14 and 24
Description: The HAQ health scale is a measure of overall health. Participants are asked to rate how well they are doing on a scale of 0 to 100, where zero represents very well and 100 represents very poor health.
Time Frame: Baseline, Week 14, Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pegloticase Plus Methotrexate
Number analyzed (Participants) | 11
score on a scale
  Change at Week 14: number analyzed (Participants) | 6
  Change at Week 14 | 8.00 (45.343)
  Change at Week 24: number analyzed (Participants) | 5
  Change at Week 24 | -11.40 (24.389)

ADVERSE EVENTS:
Time Frame: From enrollment (all-cause mortality) or first dose of study drug (adverse events) up to Week 48 + 30 days (±3 days)
Groups:
- MTX Run-In Period: MTX 15 or 25 mg SC weekly during the 6-week MTX Run-in Period.
- Pegloticase + MTX Treatment Period: Pegloticase 8 mg IV every 2 weeks and MTX 15 or 25 mg SC weekly for up to 24 weeks during the treatment period. Participants may opt to receive pegloticase with MTX for an additional 24 weeks.
Arm/Group | MTX Run-In Period | Pegloticase + MTX Treatment Period
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/13 | 1/11
Other Adverse Events (participants affected / at risk) | 7/13 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MTX Run-In Period (N=13) | Pegloticase + MTX Treatment Period (N=11)
Perineal abscess (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MTX Run-In Period (N=13) | Pegloticase + MTX Treatment Period (N=11)
Angina pectoris (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
Injection site bruising (General disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Blood glucose increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 6 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any investigator/institution that plans on presenting/publishing results provide written notification of their request 60 days prior to their presentation/publication. Horizon requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Horizon needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT04772313/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT04772313/SAP_001.pdf